CLINICAL TRIAL: NCT01644513
Title: Evaluation of Genetic Variants in Patients Under Treatment for Choroidal Neovascular (CNV) Age-related Macular Degeneration (AMD), Receiving Intravitreal Anti-VEGF Injections (Bevacizumab or Ranibizumab) to Evaluate the Association Between Genetic Load and Response to Therapy/Treatment Burden
Brief Title: Evaluation of the Association Between Genetic Load and Response to Anti-VEGF Therapy in AMD Patients
Acronym: EVERGREEN
Status: Completed | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Collaborators: Center for Eye Research and Education (Unknown)
Responsible Party: Sponsor
Other Study IDs: SCMM-AMD-105
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2012-07

CONDITIONS: Age Related Macular Degeneration
Keywords: Age Related Macular Degeneration; Choroidal Neovascular; anti-VEGF Therapy
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Remnant samples of DNA will be destroyed after analysis is complete.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Positive Responders: Have received at least one injection with no evidence of residual subretinal or intra-retinal fluid present on Spectral Domain Optical Coherence Tomography (SDOCT) one month (+/- 1 week) following most recent injection.
- Suboptimal Responders: Have received three or more injections in last six months with residual subretinal or intra-retinal fluid present on SDOCT one month (+/- 1 week) following most recent injection; Have not demonstrated complete resolution of fluid following any of the injections in the last 6 months Show leakage on Fluorescein Angiography (FA) or Indocyanine Green (ICG) imaging at some time during last 12 months

SUMMARY:
Patients with AMD who are being or have been treated with eye injections of drugs known as anti-VEGF agents with either good or poor response will have DNA collected with check swabs for analysis.

DETAILED DESCRIPTION:
The study is designed as a single-center, observational case control evaluation to compare the genetic profiles of two groups of patients categorized according to anti-VEGF treatment response as either "positive" or "suboptimal" responders following treatment with either bevacizumab or ranibizumab anti-VEGF agents. Positive and suboptimal responders will be compared to determine if genetic variant distribution or total genetic load is associated with anti-VEGF treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female 55 years of age and older
* Subject is self-reported as non-Hispanic Caucasian
* Subject provides a signed and dated informed consent
* Subject agrees to provide two buccal swabs in accordance with this protocol
* Diagnosis of CNV secondary to AMD in at least one eye
* Subject satisfies one of the following:

  1. Has received at least one injection of anti-VEGF therapy (bevacizumab or ranibizumab) with no evidence of residual subretinal or intra-retinal fluid present on SDOCT one month (+/- 1 week) following most recent injection; or
  2. Has received three or more injections in last six months with residual subretinal or intra-retinal fluid present on SDOCT one month (+/- 1 week) following most recent injection, has not shown complete resolution of fluid following any injection in last 6 months, and shows leakage on FA or ICG imaging at some time during last 12 months.

Exclusion Criteria:

* Previous sample donation under this protocol
* Presence of retinal disease involving the photoreceptors and/or outer retinal layers other than AMD loss such as high myopia, retinal dystrophies, central serous retinopathy, vein occlusion, diabetic retinopathy and uveitis or similar outer retinal diseases which have been present prior to the age of 50.
* Opacities of the ocular media, limitations of pupillary dilation or other problems sufficient to preclude adequate imaging of the posterior segment.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with age-related macular degeneration treated with anti-VEGF therapy
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Consultants Boston, Boston, Massachusetts, United States